CLINICAL TRIAL: NCT06164938
Title: Study of Cerebral Glucose Metabolism in Healthy Volunteers Using 18 F-FDG PET: Evaluation of the Effects of Aging, Comparative Evaluation of Neurodegenerative and Psychiatric Pathologies.
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: FDG-NORM
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Neuro-Degenerative Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic accuracy — The aim is to obtain a regional measure of brain glucose metabolism in each normal subject because this is a functional measure of brain activity.

SUMMARY:
The aim of the study is to obtain information on cerebral glucose metabolism measured with the 18F-FDG PET technique in normal subjects without current or previous neurological or psychiatric pathologies in order to use the data obtained for voxel-based statistical analyzes for comparison with individual subjects ( patients with disease neurological or psychiatric) which will be evaluated with the same method to improve the specificity and diagnostic sensitivity of the FDG PET exam.

The objective is to obtain a functional measure of brain glucose metabolism in every normal subject because this is a functional measure of brain activity. The subjects will represent different decades of age to have a wider range of comparison with patients.

ELIGIBILITY:
Inclusion Criteria:

* absence of neurological and psychiatric pathologies, negative pregnancy test.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 healthy volunteers, over 40 years of age, capable of understanding and wanting, who have not had a previous clinical history of neurological or psychiatric diseases, will be enrolled. Subjects with cognitive impairment and who at the time of recruitment are taking drugs active on the central nervous system will be excluded.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2010-04-14 (Actual); Primary Completion 2011-01-12 (Actual); Study Completion 2011-01-12 (Actual)

PRIMARY OUTCOMES:
Study of glucose metabolism with 18 F FDG PET | 1 year
  Study of glucose metabolism with 18 F FDG PET in normal subjects without current or previous neurological or psychiatric pathologies in order to use the data obtained for statistical analyzes for comparison with individual subjects (patients with neurological or psychiatric) which will be evaluated with the same method to improve the diagnostic sensitivity of the FDG PET exam.

IPD SHARING:
Plan to Share IPD: No